CLINICAL TRIAL: NCT01214083
Title: N-acetylcysteine Plus Naltrexone for the Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDA-2-014-09F
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Alcoholism
Keywords: N-acetylcysteine; naltrexone
MeSH Terms: conditions — Alcoholism | interventions — Acetylcysteine; Naltrexone; Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): N-acetylcysteine + high-dose naltrexone (150 mg)
  Interventions: Drug: N-acetylcysteine + high-dose naltrexone (150 mg)
- Arm 2 (Experimental): High-dose naltrexone (150 mg) alone
  Interventions: Drug: High-dose naltrexone (150 mg) alone
- Arm 3 (Active Comparator): Low-dose naltrexone (50 mg) alone
  Interventions: Drug: Low-dose naltrexone (50 mg) alone

INTERVENTIONS:
Drug: N-acetylcysteine + high-dose naltrexone (150 mg) — All subjects will be evaluated weekly for 12 weeks.
  Arms: Arm 1
Drug: High-dose naltrexone (150 mg) alone — All subjects will be evaluated weekly for 12 weeks.
  Arms: Arm 2
Drug: Low-dose naltrexone (50 mg) alone — All subjects will be evaluated weekly for 12 weeks.
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine whether: (1) the combination of N-acetylcysteine + high-dose naltrexone (150 mg) works better than high-dose naltrexone (150 mg) alone in reducing alcohol drinking; and (2) high-dose naltrexone (150 mg) alone works better than low-dose naltrexone (50 mg) alone in reducing alcohol drinking.

DETAILED DESCRIPTION:
The 3 groups (N-acetylcysteine plus naltrexone 150 mg, naltrexone 150 mg, and naltrexone 50 mg) will be compared in a 12-week randomized, double-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* alcohol dependence by DSM-IV criteria
* heavy drinking at least 6 times within the past month ('heavy drinking' defined as 5 or more standard drinks per day for men and 4 or more standard drinks for women)
* able to provide informed consent
* a score of 6 or more on the Penn Alcohol Craving Scale (PACS)
* subject agrees not to take over-the-counter analgesics during the study

Exclusion Criteria:

* current drug abuse or dependence by DSM-IV criteria (except nicotine and marijuana)
* current psychotic disorders or bipolar disorders
* current suicidal or homicidal ideation
* positive illicit drug screen test (except marijuana)
* ongoing narcotic use or risks for narcotic use during the study
* increased risk for severe alcohol withdrawal by a score of 10 or more on the Clinical Institute Withdrawal Assessment for Alcohol, Revised (CIWA-Ar)
* clinically significant cardiac, hepatic, renal, neurologic, or pulmonary disease
* baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3 times normal
* current use of disulfiram, acamprosate or topiramate
* pregnant or nursing, or inadequate birth control methods in women of childbearing potential
* alcohol breathalyzer level 0.08 or more at the screening visit
* severe alcohol withdrawal (delirium tremens or withdrawal seizures) within the past year
* currently requiring inpatient treatment for treating alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-10-15 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 111 subjects signed consent. Of 111 subjects, 95 subjects were qualified for the trial.
Period: Overall Study
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Started | 31 | 33 | 31
Completed | 19 | 23 | 21
Not Completed | 12 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone | Total
Number analyzed (Participants) | 31 | 33 | 31 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 33 | 31 | 95
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 29 | 28 | 29 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 33 | 31 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days
Description: "Percentage of heavy drinking days" was measured by the Time Line Follow Back (TLFB) Method. ('Heavy drinking' was defined as 5 or more standard drinks per day for men and 4 or more standard drinks for women.) The percentage has a total range of 0%-100%. Higher percentages represent a worse outcome (i.e., more heavy drinking).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
percentage of heavy drinking days
  Percentage of heavy drinking days at week 1 | 45.0 (4.5) | 50.6 (4.3) | 44.0 (4.5)
  Percentage of heavy drinking days at week 13 | 5.2 (5.6) | 3.4 (5.1) | 3.3 (5.3)

2. Secondary Outcome: Liver Function Tests (AST)
Time Frame: week 0 and week 13
Measure: Mean (Standard Error); unit: units/liter
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units/liter
  Liver function tests (AST) at week 0 | 34.7 (6.6) | 29.0 (6.4) | 30.0 (6.6)
  Liver function tests (AST) at week 13 | 27.3 (7.9) | 32.1 (7.4) | 22.2 (7.5)

3. Secondary Outcome: Penn Alcohol Craving Scale (PACS)
Description: The Penn Alcohol Craving Scale is designed to assess alcohol craving severity. The scale has a total score range of 0-30. Higher values represent a worse outcome (i.e., higher craving).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units on a scale
  Penn Alcohol Craving Scale at week 1 | 18.0 (1.1) | 18.4 (1.1) | 16.1 (1.1)
  Penn Alcohol Craving Scale at week 13 | 7.2 (1.4) | 8.3 (1.3) | 6.3 (1.3)

4. Secondary Outcome: Obsessive Compulsive Drinking Scale (OCDS)
Description: The Obsessive Compulsive Drinking Scale is designed to assess obsessive and compulsive aspects of alcoholism. The scale has a total score range of 0-56. Higher values represent a worse outcome (i.e., more alcohol problems).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units on a scale
  Obsessive Compulsive Drinking Scale at week 1 | 28.2 (1.8) | 29.0 (1.7) | 24.5 (1.8)
  Obsessive Compulsive Drinking Scale at week 13 | 9.1 (2.1) | 14.0 (1.9) | 9.0 (2.0)

5. Secondary Outcome: Clinical Global Impression (CGI)
Description: The Clinical Global Impression is designed to assess overall severity of illness. The scale has a total score range of 1-7. Higher values represent a worse outcome (i.e., severe illness).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units on a scale
  Clinical Global Impression at week 1 | 3.7 (0.1) | 3.7 (0.1) | 3.6 (0.1)
  Clinical Global Impression at week 13 | 1.5 (0.2) | 1.7 (0.2) | 1.4 (0.2)

6. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire is designed to assess a quality of life. The scale has a total score range of 16-80. Higher values represent a better outcome (i.e., better quality of life).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units on a scale
  Q-LES-Q at week 1 | 53.2 (1.9) | 53.8 (1.8) | 55.1 (1.9)
  Q-LES-Q at week 13 | 61.6 (2.1) | 59.6 (2.0) | 63.9 (2.1)

7. Secondary Outcome: Percentage of Drinking Days
Description: "Percentage of drinking days" was measured by the Time Line Follow Back (TLFB) Method. The percentage has a total range of 0%-100%. Higher percentages represent a worse outcome (i.e., more drinking days).
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: percentage of drinking days
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
percentage of drinking days
  percentage of drinking days at week 1 | 64.6 (6.3) | 63.8 (6.1) | 55.3 (6.3)
  percentage of drinking days at week 13 | 21.1 (7.6) | 24.5 (7.0) | 18.2 (7.3)

8. Secondary Outcome: Drinks Per Drinking Days
Time Frame: week 1 and week 13
Measure: Mean (Standard Error); unit: drinks/drinking day
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
drinks/drinking day
  drinks per drinking days at week 1 | 7.3 (0.6) | 5.9 (0.6) | 7.3 (0.6)
  drinks per drinking days at week 13 | 1.1 (0.6) | 1.2 (0.6) | 1.0 (0.6)

9. Secondary Outcome: Liver Function Tests (ALT)
Time Frame: week 0 and week 13
Measure: Mean (Standard Error); unit: units/liter
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Number analyzed (Participants) | 31 | 33 | 31
units/liter
  Liver Function Tests (ALT) at week 0 | 49.4 (12.0) | 36.5 (11.6) | 34.7 (12.0)
  Liver Function Tests (ALT) at week 13 | 27.6 (13.9) | 40.1 (13.0) | 31.3 (13.2)

ADVERSE EVENTS:
Arm/Group | N-acetylcysteine + High-dose Naltrexone (150 mg) | High-dose Naltrexone (150 mg) Alone | Low-dose Naltrexone (50 mg) Alone
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 14/31 | 12/33 | 9/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine + High-dose Naltrexone (150 mg) (N=31) | High-dose Naltrexone (150 mg) Alone (N=33) | Low-dose Naltrexone (50 mg) Alone (N=31)
Nausea (Gastrointestinal disorders) | 9 | 9 | 5
Drowsiness (General disorders) | 1 | 4 | 0
Headache (General disorders) | 3 | 1 | 2
Decreased appetite (General disorders) | 2 | 1 | 2
Dry mouth (General disorders) | 2 | 2 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No